CLINICAL TRIAL: NCT04610892
Title: A Phase IIB, Randomized, Double Blinded, Placebo Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of MEDI6570 in Participants With a Prior Myocardial Infarction and Persistent Inflammation
Brief Title: Efficacy and Safety of MEDI6570 in Patients With a History of Myocardial Infarction
Acronym: GOLDILOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: The TIMI Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4920C00002; 2020-000840-75 (EudraCT Number)
Record Dates: First submitted 2020-07-28; First posted 2020-11-02 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Coronary Heart Disease (CHD)
Keywords: Coronary Heart Disease; Atherosclerosis
MeSH Terms: conditions — Coronary Disease; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- MEDI6570 Low dose (Experimental): Monthly Subcutaneous administration.
  Interventions: Biological: MEDI6570
- MEDI6570 Medium dose (Experimental): Monthly Subcutaneous administration.
  Interventions: Biological: MEDI6570
- MEDI6570 High dose (Experimental): Monthly Subcutaneous administration.
  Interventions: Biological: MEDI6570
- Placebo Low dose (Placebo Comparator): Monthly Subcutaneous administration.
  Interventions: Biological: Placebo
- Placebo Medium dose (Placebo Comparator): Monthly Subcutaneous administration
  Interventions: Biological: Placebo
- Placebo High dose (Placebo Comparator): Monthly Subcutaneous administration
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MEDI6570 — MEDI6570
  Arms: MEDI6570 High dose; MEDI6570 Low dose; MEDI6570 Medium dose
Biological: Placebo — Buffer
  Arms: Placebo High dose; Placebo Low dose; Placebo Medium dose

SUMMARY:
A Phase IIB Parallel group Study to Evaluate the Efficacy and Safety of MEDI6570 in Participants with a Prior Myocardial Infarction.

DETAILED DESCRIPTION:
This Phase IIB, proof-of-concept, dose-range finding clinical study is being conducted to evaluate the anti-inflammatory potential of MEDI6570 and its effect on surrogates for atherosclerotic and heart failure (HF) events in patients with a history of myocardial infarction (MI). The results of the Phase IIB study will inform future clinical development options and precision medicine strategy for future clinical studies.

Participants will be randomized in a 2:2:1:1 ratio after protocol Amend 2, 360 evaluable participants (111 evaluable participants in each of the 2 MEDI6570 groups, plus 27 evaluable participants in the legacy low dose MEDI6570 group, plus 111 participants in pooled placebo) will complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must provide informed consent before any study specific activities are performed, must be able and willing to meet all requirements for randomization within 42 days after signing the full ICF, and must adhere to the schedules of activities.
2. Women must be ≥ 40 years of age at the time of signing the ICF. Men must be ≥ 21 years of age at the time of signing the ICF.
3. Participant must:

   1. be 30 to 365 days after presumed type-1 (ie, due to plaque rupture or erosion) MI (either STEMI or NSTEMI) at the time of enrollment.
   2. have persistent inflammation, defined as hs CRP ≥ 1 mg/L, as measured centrally at screening Visit 1.
4. Participant must have body mass index within the range 18 to 40 kg/m2 inclusive.
5. For female participants, the participant must not be pregnant or lactating and must be of non-childbearing potential, confirmed at screening Visit 1 by one of the following:

   1. Postmenopausal, defined as amenorrhea for ≥ 12 months following cessation of all exogenous hormonal treatments, and with luteinizing hormone and follicle stimulating hormone levels in the postmenopausal range.
   2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy. Tubal ligation is not considered as irreversible surgical sterilization.
6. Participant must have an evaluable, pre-randomization CTA with quantifiable, non calcified plaque.

Exclusion Criteria:

1. History of any clinically important disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
2. Percutaneous coronary intervention or diagnostic angiogram planned after screening. Eligible participants who have a diagnostic angiogram performed in the absence of undergoing a new PCI may continue screening after the diagnostic angiogram has been performed or may be rescreened.
3. History of or planned coronary artery bypass grafting.
4. Documented episode of post-MI pericarditis in the 3 months before enrollment.
5. Ongoing New York Heart Association Class IV HF.
6. Increased risk of bleeding

   1. Patients with history or presence of any bleeding disorder.
   2. Signs of ongoing bleeding at screening (eg, identified macroscopic bleeding, low hemoglobin presumed to be caused by bleeding) or high risk for major bleeding in accordance with the Investigator's assessment.
   3. Need for chronic therapeutic anticoagulation therapy anticipated to be required throughout the course of the study (short-term treatment with prophylactic doses of heparin/low molecular weight heparin are allowed).
   4. Known severe liver disease.
7. History or presence of any of the following:

   1. Ongoing infection or febrile illness that in the opinion of the investigator may be the cause of elevated hs-CRP on screening.
   2. Ongoing atrial fibrillation or flutter.
   3. Cancer within 5 years before randomization, with the exception of non melanoma skin cancer.
   4. Alcohol or substance abuse within 6 months before randomization, as judged by the investigator.
   5. Known history of hypersensitivity reactions to other biologics, to human IgG preparations, or to any component of MEDI6570, or ongoing severe allergy as judged by the investigator.
   6. Patients with active positive results on screening for serum hepatitis B surface antigen, hepatitis C antibody, or HIV.
8. Any clinically important abnormalities in clinical chemistry, hematology, coagulation parameters, as judged by the investigator.
9. BP values at screening:

   1. Systolic BP < 90 mmHg or > 180 mmHg.
   2. Diastolic BP > 100 mmHg.
   3. Participants who are excluded based on elevated BP may be rescreened following adequate treatment.
10. Participants with any of the following contraindications to CTA:

    1. eGFR < 50 mL/min/1.73 m2 by the Chronic Kidney Disease Epidemiology Collaboration equation, or end stage renal disease treated with kidney transplant or renal replacement therapy.
    2. Allergy to iodinated contrast.
    3. History of contrast-induced nephropathy.
    4. Contraindication to nitroglycerin.
    5. Rapid heart rate that is uncontrolled by medical therapy.
    6. Inability to hold breath for at least 6 seconds.
11. Receipt of any investigational device or therapy within 6 months or 5 half lives before screening (whichever is longer).

    This criterion does NOT apply for inactive, non replicating COVID-19 vaccines approved by Health Authorities or under emergency use authorization.
12. Planned participation in an additional investigational study of an intervention or biologic before the end of the follow-up period. Participation in observational studies or studies without investigational drugs or devices is allowed.
13. Participants who are legally institutionalized.
14. An employee or close relative of an employee of the sponsor, the CRO, or the study site, regardless of the employee or close relative's role.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (77):
- United States (18):
  - Research Site, Mobile, Alabama
  - Research Site, Beverly Hills, California
  - Research Site, Covina, California
  - Research Site, Northridge, California
  - Research Site, Torrance, California
  - Research Site, Ponte Vedra, Florida
  - Research Site, Decatur, Georgia
  - Research Site, Muncie, Indiana
  - Research Site, Richmond, Indiana
  - Research Site, West Des Moines, Iowa
  - Research Site, Midland, Michigan
  - Research Site, Columbia, Missouri
  - Research Site, New Brunswick, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, Canton, Ohio
  - Research Site, Rapid City, South Dakota
  - Research Site, Winchester, Virginia
  - Research Site, Madison, Wisconsin
- Australia (5):
  - Research Site, Adelaide
  - Research Site, Bedford Park
  - Research Site, Clayton
  - Research Site, Murdoch
  - Research Site, Perth
- Canada (3):
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Czechia (6):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Liberec
  - Research Site, Pardubice
  - Research Site, Plzen - Bory
  - Research Site, Prague
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Székesfehérvár
- Italy (4):
  - Research Site, Cona
  - Research Site, Milan
  - Research Site, Parma
  - Research Site, Rozzano
- Japan (12):
  - Research Site, Himeji-shi
  - Research Site, Kasuga-shi
  - Research Site, Kasugai-shi
  - Research Site, Kitakyushu-shi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Matsudo-Shi
  - Research Site, Minamiku
  - Research Site, Miyazaki
  - Research Site, Morioka
  - Research Site, Osaka
  - Research Site, Sendai
- Netherlands (8):
  - Research Site, Alkmaar
  - Research Site, Deventer
  - Research Site, Heerlen
  - Research Site, Nijmegen
  - Research Site, Tilburg
  - Research Site, Utrecht
  - Research Site, Venlo
  - Research Site, Zwolle
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Opole
  - Research Site, Wroclaw
- Spain (7):
  - Research Site, Barcelona
  - Research Site, El Palmar
  - Research Site, Hospitalet de Llobregat(Barcel
  - Research Site, Madrid
  - Research Site, Pontevedra
  - Research Site, Santiago de Compostela
  - Research Site, Seville
- United Kingdom (5):
  - Research Site, Aylesbury
  - Research Site, Exeter
  - Research Site, Middlesbrough
  - Research Site, Newcastle upon Tyne
  - Research Site, Wythenshawe

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4920C00002&attachmentIdentifier=596f3ac2-1432-4b10-b785-8bf7e7a911d6&fileName=D4920C00002_redacted_CSP.pdf&versionIdentifier=
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4920C00002&attachmentIdentifier=7c8d42e1-7892-43fd-85de-c2dbbcd00c67&fileName=D4920C00002_redacted_SAP.pdf&versionIdentifier=
- See also: redacted CSR — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4920C00002&attachmentIdentifier=4135a31f-bf26-4a01-bd9c-fda516aec2ef&fileName=D4920C00002-_redacted_CSR_synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- MEDI6570 50 mg: Participants received MEDI6570 50 mg every 4 weeks for 32 weeks
- MEDI6570 150 mg: Participants received MEDI6570 150 mg every 4 weeks for 32 weeks
- MEDI6570 250 mg/400 mg: Participants received MEDI6570 250 mg/400 mg every 4 weeks for 32 weeks.
- MEDI6570 400 mg: Participants received MEDI6570 400 mg every 4 weeks for 32 weeks
- Placebo: Participants received Placebo matched to MEDI6570 every 4 weeks for 32 weeks
Period: Overall Study
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 250 mg/400 mg | MEDI6570 400 mg | Placebo
Started | 40 | 129 | 8 (MEDI6570 250 mg/400 mg : subjects initially randomized to 250 mg that switched dose to 400 mg during the trial.) | 118 | 128
Completed | 35 | 126 | 8 | 110 | 117
Not Completed | 5 | 3 | 0 | 8 | 11
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 3
Not completed — Death | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 0 | 6 | 6
Not completed — Subjects who did not receive treatment | 1 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: 8 subjects initially randomized to the 250 mg group switched dose to 400 mg following CSP amendment 1 and were analysed according to the 400 mg group.
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | Placebo | Total
Number analyzed (Participants) | 40 | 129 | 126 | 128 | 423
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (8.3) | 59.9 (9.2) | 59.4 (9.6) | 60.4 (9.5) | 59.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 19 | 23 | 21 | 75
  Male | 28 | 110 | 103 | 107 | 348
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 2 | 7 | 19
  Not Hispanic or Latino | 35 | 124 | 124 | 121 | 404
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 0 | 1 | 1
  ASIAN | 7 | 10 | 8 | 9 | 34
  BLACK OR AFRICAN AMERICAN | 0 | 1 | 0 | 0 | 1
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 1 | 0 | 0 | 1
  OTHER | 0 | 1 | 0 | 0 | 1
  WHITE | 33 | 116 | 118 | 118 | 385
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 33 | 116 | 118 | 118 | 385
  Non-caucasian | 7 | 13 | 8 | 10 | 38
  Missing | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  Australia | 0 | 6 | 6 | 3 | 15
  Canada | 0 | 3 | 1 | 0 | 4
  Czech Republic | 2 | 17 | 17 | 18 | 54
  Hungary | 9 | 11 | 12 | 23 | 55
  Italy | 0 | 14 | 21 | 19 | 54
  Japan | 7 | 9 | 8 | 8 | 32
  Netherlands | 1 | 18 | 11 | 11 | 41
  Poland | 2 | 14 | 14 | 10 | 40
  Spain | 13 | 20 | 18 | 18 | 69
  United Kingdom | 0 | 5 | 5 | 1 | 11
  United States of America | 6 | 12 | 13 | 17 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 253 in Non-calcified Plaque Volume in the Most Diseased Coronary Segment (NCPVMD), as Measured by Computed Tomography Angiography (CTA) Imaging
Description: To evaluate the effect of MEDI6570 on non-calcified coronary atherosclerotic plaques compared with placebo. The primary endpoint of change in NCPVMD from baseline to Day 253 was assessed based on the CTA Analysis Populations.
Time Frame: From baseline to Day 253
Population: Participants within the Intention To Treat (ITT) Population who had interpretable CTA scans at baseline and at Day 253. Participants were analyzed according to their randomized treatment group.
  Subjects initially randomized to the 250 mg group switched dose to 400 mg following clinical study protocol (CSP) amendment 1 and were analysed according to the 400 mg group.
Measure: Least Squares Mean (Standard Error); unit: mm^3
Groups:
- MEDI6570 150 mg or 400 mg: Participants received MEDI6570 150 mg or 400 mg every 4 weeks for 32 weeks
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | MEDI6570 150 mg or 400 mg | Placebo
Number analyzed (Participants) | 35 | 127 | 118 | 245 | 117
mm^3 | -15.3220 (4.9219) | -4.5509 (3.1654) | -6.3658 (3.2559) | -5.4220 (2.6622) | -6.9424 (3.2729)
Statistical Analysis 1: Comparison: MEDI6570 50 mg vs Placebo; Test type: Superiority; p = 0.065, ANCOVA — One-sided p-value; The treatment as a fixed effects and the baseline value and the geographic region and statin therapy intensity at screening as covariates; Least Square Mean difference = -8.3797, 90% CI [-17.4980 to 0.7387]
Statistical Analysis 2: Comparison: MEDI6570 150 mg vs Placebo; Test type: Superiority; p = 0.747, ANCOVA — One-sided p-value; [statistical method as in outcome 1, analysis 1]; Least Square Mean difference = 2.3915, 90% CI [-3.5338 to 8.3167]
Statistical Analysis 3: Comparison: MEDI6570 400 mg vs Placebo; Test type: Superiority; p = 0.563, ANCOVA — One-sided p-value; [statistical method as in outcome 1, analysis 1]; Least Square Mean difference = 0.5766, 90% CI [-5.4389 to 6.5921]
Statistical Analysis 4: Comparison: MEDI6570 150 mg or 400 mg vs Placebo; Test type: Superiority; p = 0.685, ANCOVA — One-sided p-value; [statistical method as in outcome 1, analysis 1]; Least Square Mean difference = 1.5204, 90% CI [-3.6657 to 6.7064]

2. Secondary Outcome: Change From Baseline to Day 253 in N Terminal Prohormone Brain Natriuretic Peptide (NT-proBNP)
Description: To evaluate the effect of MEDI6570 on a surrogate biomarker of Heart Failure (HF) compared with placebo
Time Frame: From baseline to Day 253
Population: Randomized subjects who received any study treatment will be included in the As-treated Population. Subjects will be analysed according to the actual treatment they received, regardless of their randomized treatment group. Subjects treated within 250 mg group that received at least one 400 mg dose during the study will be analysed according to the 400mg group.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | MEDI6570 150 mg or 400 mg | Placebo
Number analyzed (Participants) | 35 | 125 | 123 | 248 | 118
pg/mL | 0.8226 (9.4) | 0.7787 (5.5) | 0.7368 (5.6) | 0.7575 (4.4) | 0.7370 (5.6)
Statistical Analysis 1: Comparison: MEDI6570 50 mg vs Placebo; Test type: Superiority; p = 0.854, Mixed model with repeated measurements — One sided p-value; The model was adjusted for the baseline value and the stratification factors (geographic region and statin therapy intensity at screening); Geometric LS mean ratio estimate = 1.12, 90% CI [0.94 to 1.33]
Statistical Analysis 2: Comparison: MEDI6570 150 mg vs Placebo; Test type: Superiority; p = 0.790, Mixed model with repeated measurements — One sided p-value; [statistical method as in outcome 2, analysis 1]; Geometric LS mean ratio estimate = 1.06, 90% CI [0.94 to 1.18]
Statistical Analysis 3: Comparison: MEDI6570 400 mg vs Placebo; Test type: Superiority; p = 0.498, Mixed model with repeated measurements — One sided p-value; [statistical method as in outcome 2, analysis 1]; Geometric LS mean ratio estimate = 1.00, 90% CI [0.89 to 1.12]
Statistical Analysis 4: Comparison: MEDI6570 150 mg or 400 mg vs Placebo; Test type: Superiority; p = 0.678, Mixed model with repeated measurements — One sided p-value; [statistical method as in outcome 2, analysis 1]; Geometric LS mean ratio estimate = 1.03, 90% CI [0.93 to 1.13]

3. Secondary Outcome: Change From Baseline to Day 253 in Left Ventricular Ejection Fraction (LVEF)
Description: To evaluate the effect of MEDI6570 on left ventricular systolic function compared with placebo
Time Frame: From baseline to Day 253
Population: Subjects within the ITT population who have interpretable echocardiograms in the baseline and follow-up periods will be included in the Echocardiogram Analysis Population. Subjects will be analysed according to their randomized treatment group. subjects initially randomized to the 250 mg group switched dose to 400 mg following CSP amendment 1 and were analysed according to the 400 mg group
Measure: Least Squares Mean (Standard Error); unit: Percentage of LVEF
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | MEDI6570 150 mg or 400 mg | Placebo
Number analyzed (Participants) | 31 | 115 | 112 | 227 | 103
Percentage of LVEF | -0.91 (0.55) | 0.32 (0.34) | 0.11 (0.35) | 0.22 (0.28) | 0.53 (0.35)
Statistical Analysis 1: Comparison: MEDI6570 50 mg vs Placebo; Test type: Superiority; p = 0.990, ANCOVA — One sided p-value; The model was adjusted for the baseline value and stratification factors (geographic region and statin therapy intensity at screening); Least Squares mean difference = -1.44, 90% CI [-2.44 to -0.43]
Statistical Analysis 2: Comparison: MEDI6570 150 mg vs Placebo; Test type: Superiority; p = 0.697, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -0.21, 90% CI [-0.87 to 0.45]
Statistical Analysis 3: Comparison: MEDI6570 400 mg vs Placebo; Test type: Superiority; p = 0.849, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -0.42, 90% CI [-1.08 to 0.25]
Statistical Analysis 4: Comparison: MEDI6570 150 mg or 400 mg vs Placebo; Test type: Superiority; p = 0.811, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -0.31, 90% CI [-0.89 to 0.27]

4. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF) Change From Baseline to Day 253 Among Subjects With Reduced Ejection Fraction (< 50%)
Description: To evaluate the effect of MEDI6570 on left ventricular systolic function among participants with reduced ejection fraction (defined as <50%) compared with placebo
Time Frame: From baseline to Day 253
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percentage of LVEF
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | MEDI6570 150 mg or 400 mg | Placebo
Number analyzed (Participants) | 7 | 13 | 20 | 33 | 14
Percentage of LVEF | -1.08 (1.52) | 1.32 (1.13) | 2.09 (1.00) | 1.79 (0.82) | 2.41 (1.04)
Statistical Analysis 1: Comparison: MEDI6570 50 mg vs Placebo; Test type: Superiority; p = 0.972, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -3.50, 90% CI [-6.49 to -0.50]
Statistical Analysis 2: Comparison: MEDI6570 150 mg vs Placebo; Test type: Superiority; p = 0.777, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -1.10, 90% CI [-3.49 to 1.30]
Statistical Analysis 3: Comparison: MEDI6570 400 mg vs Placebo; Test type: Superiority; p = 0.596, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -0.32, 90% CI [-2.54 to 1.89]
Statistical Analysis 4: Comparison: MEDI6570 150 mg or 400 mg vs Placebo; Test type: Superiority; p = 0.698, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -0.63, 90% CI [-2.64 to 1.38]

5. Secondary Outcome: Change From Baseline to Day 253 in Global Longitudinal Strain (GLS)
Description: To evaluate the effect of MEDI6570 on left ventricular systolic function compared with placebo
Time Frame: From baseline to Day 253
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percentage of GLS
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | MEDI6570 150 mg or 400 mg | Placebo
Number analyzed (Participants) | 29 | 105 | 109 | 214 | 100
Percentage of GLS | -1.20 (0.56) | -0.70 (0.35) | -0.77 (0.35) | -0.74 (0.29) | 0.09 (0.35)
Statistical Analysis 1: Comparison: MEDI6570 50 mg vs Placebo; Test type: Superiority; p = 0.981, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -1.29, 90% CI [-2.32 to -0.27]
Statistical Analysis 2: Comparison: MEDI6570 150 mg vs Placebo; Test type: Superiority; p = 0.974, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -0.80, 90% CI [-1.47 to -0.12]
Statistical Analysis 3: Comparison: MEDI6570 400 mg vs Placebo; Test type: Superiority; p = 0.983, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -0.86, 90% CI [-1.53 to -0.20]
Statistical Analysis 4: Comparison: MEDI6570 150 mg or 400 mg vs Placebo; Test type: Superiority; p = 0.990, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -0.83, 90% CI [-1.42 to -0.25]

6. Secondary Outcome: Global Longitudinal Strain (GLS) Change From Baseline to Day 253 Among Subjects With Reduced Ejection Fraction (< 50%)
Description: as for outcome 4
Time Frame: From baseline to Day 253
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percentage of GLS
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | MEDI6570 150 mg or 400 mg | Placebo
Number analyzed (Participants) | 6 | 12 | 20 | 32 | 15
Percentage of GLS | -0.39 (1.03) | -1.16 (0.78) | 0.41 (0.64) | -0.19 (0.55) | 1.76 (0.66)
Statistical Analysis 1: Comparison: MEDI6570 50 mg vs Placebo; Test type: Superiority; p = 0.959, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -2.14, 90% CI [-4.16 to -0.12]
Statistical Analysis 2: Comparison: MEDI6570 150 mg vs Placebo; Test type: Superiority; p = 0.998, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -2.92, 90% CI [-4.53 to -1.31]
Statistical Analysis 3: Comparison: MEDI6570 400 mg vs Placebo; Test type: Superiority; p = 0.939, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -1.35, 90% CI [-2.79 to 0.09]
Statistical Analysis 4: Comparison: MEDI6570 150 mg or 400 mg vs Placebo; Test type: Superiority; p = 0.991, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -1.94, 90% CI [-3.27 to -0.62]

7. Secondary Outcome: Change From Baseline to Day 253 in Global Non-calcified Plaque Volume (NCPV)
Description: To evaluate the effect of MEDI6570 on other measures of non-calcified coronary atherosclerotic plaque compared with placebo
Time Frame: From baseline to Day 253
Population: Participants within the ITT Population who had interpretable b CTA scans at baseline and at Day 253 or at Day 122 were included. (Note that separate analyses were conducted for Day 253 and Day 122). Participants were analyzed according to their randomized treatment group.
  Subjects initially randomized to the 250 mg group switched dose to 400 mg following CSP amendment 1 and were analysed according to the 400 mg group.
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | MEDI6570 150 mg or 400 mg | Placebo
Number analyzed (Participants) | 34 | 125 | 116 | 241 | 117
mm^3 | -26.4453 (10.0524) | -10.9010 (6.4671) | -10.4850 (6.6607) | -10.7013 (5.4415) | -10.3083 (6.7052)
Statistical Analysis 1: Comparison: MEDI6570 50 mg vs Placebo; Test type: Superiority; p = 0.077, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -16.1370, 90% CI [-34.7829 to 2.5089]
Statistical Analysis 2: Comparison: MEDI6570 150 mg vs Placebo; Test type: Superiority; p = 0.468, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -0.5927, 90% CI [-12.7267 to 11.5413]
Statistical Analysis 3: Comparison: MEDI6570 400 mg vs Placebo; Test type: Superiority; p = 0.491, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -0.1767, 90% CI [-12.4678 to 12.1144]
Statistical Analysis 4: Comparison: MEDI6570 150 mg or 400 mg vs Placebo; Test type: Superiority; p = 0.476, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -0.3930, 90% CI [-11.0022 to 10.2162]

8. Secondary Outcome: Change From Baseline to Day 253 in Low Attenuation Plaque Volume (LAPV)
Description: as for outcome 7
Time Frame: From baseline to Day 253
Population: Participants within the ITT Population who had interpretable CTA scans at baseline and at Day 253. Participants were analyzed according to their randomized treatment group.
  Subjects initially randomized to the 250 mg group switched dose to 400 mg following CSP amendment 1 and were analysed according to the 400 mg group.
Measure: Least Squares Mean (Standard Error); unit: mm3
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | MEDI6570 150 mg or 400 mg | Placebo
Number analyzed (Participants) | 34 | 125 | 116 | 241 | 117
mm3 | -7.9167 (3.5226) | -4.8101 (2.2690) | -4.2748 (2.3363) | -4.5532 (1.9099) | -3.5733 (2.3481)
Statistical Analysis 1: Comparison: MEDI6570 50 mg vs Placebo; Test type: Superiority; p = 0.136, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -4.3435, 90% CI [-10.8637 to 2.1768]
Statistical Analysis 2: Comparison: MEDI6570 150 mg vs Placebo; Test type: Superiority; p = 0.316, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -1.2369, 90% CI [-5.4796 to 3.0059]
Statistical Analysis 3: Comparison: MEDI6570 400 mg vs Placebo; Test type: Superiority; p = 0.394, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -0.7015, 90% CI [-5.0096 to 3.6065]
Statistical Analysis 4: Comparison: MEDI6570 150 mg or 400 mg vs Placebo; Test type: Superiority; p = 0.332, ANCOVA — One sided p-value; [statistical method as in outcome 3, analysis 1]; Least Squares mean difference = -0.9799, 90% CI [-4.6927 to 2.7329]

9. Secondary Outcome: Summary of ADA (Anti-drug Antibody) Responses During the Study
Description: To evaluate the immunogenicity of MEDI6570
Time Frame: From baseline to Day 325/405. Day 325/405: for participants who completed the study under clinical study protocol (CSP) Amendment 1 & 2, the end of study visits were Day 405 and Day 325 respectively.
Population: Subjects included in the As-treated Population who have ≥ 1 immunogenicity sample will be included in the Immunogenicity Population. Subjects will be analysed according to the actual treatment they received. Subjects initially randomized to the 250 mg group switched dose to 400 mg following CSP amendment 1 and were analysed according to the 400 mg group.
Measure: Count of Participants; unit: Participants
Groups:
- MEDI6570 50 mg: Participants received MEDI6570 50 mg very 4 weeks for 32 weeks
- MEDI6570 150 mg: Participants received MEDI6570 150 mg very 4 weeks for 32 weeks
- MEDI6570 400 mg: Participants received MEDI6570 400 mg very 4 weeks for 32 weeks
- MEDI6570 Total: Number of participants received MEDI6570 50 mg, MEDI6570 150 mg and 400 mg
- Placebo: Participants received Placebo matched to MEDI6570 very 4 weeks for 32 weeks
- Total: Overall Total
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | MEDI6570 Total | Placebo | Total
Number analyzed (Participants) | 39 | 129 | 126 | 294 | 126 | 420
Participants
  ADA (anti-drug antibody) prevalence (positive at baseline or post-baseline) | 2 | 10 | 3 | 15 | 1 | 16
  ADA (anti-drug antibody) incidence (TEADA positive): number analyzed (Participants) | 38 | 128 | 124 | 290 | 123 | 413
  ADA (anti-drug antibody) incidence (TEADA positive) | 2 | 9 | 2 | 13 | 1 | 14
  Treatment-induced ADA (anti-drug antibody) positive: number analyzed (Participants) | 38 | 128 | 124 | 290 | 123 | 413
  Treatment-induced ADA (anti-drug antibody) positive | 2 | 9 | 2 | 13 | 1 | 14
  Treatment-boosted ADA (anti-drug antibody) positive: number analyzed (Participants) | 37 | 128 | 124 | 289 | 118 | 407
  Treatment-boosted ADA (anti-drug antibody) positive | 0 | 1 | 0 | 1 | 0 | 1
  ADA (anti-drug antibody) persistently positive: number analyzed (Participants) | 37 | 128 | 124 | 289 | 118 | 407
  ADA (anti-drug antibody) persistently positive | 2 | 7 | 1 | 10 | 1 | 11

10. Secondary Outcome: Anti-drug Antibody Titre Summary by Visit
Description: To evaluate the immunogenicity of MEDI6570
Time Frame: From Baseline to Day 325/405. Day 325/405: for participants who completed the study under CSP Amendment 1 & 2, the end of study visits were Day 405 and Day 325 respectively.
Population: as for outcome 9
Measure: Median (Full Range); unit: Titer units
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | MEDI6570 Total | Placebo | Total
Number analyzed (Participants) | 39 | 129 | 126 | 294 | 126 | 420
Titer units
  Baseline: number analyzed (Participants) | 0 | 1 | 1 | 2 | 0 | 2
  Baseline |  | 80 [80 to 80] | 320 [320 to 320] | 200 [80 to 320] |  | 200 [80 to 320]
  Day 29: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 1
  Day 29 |  | 640 [640 to 640] |  | 640 [640 to 640] |  | 640 [640 to 640]
  Day 57: number analyzed (Participants) | 0 | 2 | 0 | 2 | 0 | 2
  Day 57 |  | 80 [80 to 80] |  | 80 [80 to 80] |  | 80 [80 to 80]
  Day 113: number analyzed (Participants) | 1 | 1 | 0 | 2 | 0 | 2
  Day 113 | 640 [640 to 640] | 640 [640 to 640] |  | 640 [640 to 640] |  | 640 [640 to 640]
  Day 169: number analyzed (Participants) | 1 | 2 | 0 | 3 | 0 | 3
  Day 169 | 320 [320 to 320] | 1600 [640 to 2560] |  | 640 [320 to 2560] |  | 640.0 [320 to 2560]
  Day 253: number analyzed (Participants) | 1 | 3 | 2 | 6 | 0 | 6
  Day 253 | 160 [160 to 160] | 1360 [160 to 2560] | 80 [80 to 80] | 160 [80 to 2560] |  | 160 [80 to 2560]
  Day 325/405: number analyzed (Participants) | 2 | 5 | 1 | 8 | 1 | 9
  Day 325/405 | 120.0 [80 to 160] | 320 [80 to 1280] | 80 [80 to 80] | 160 [80 to 1280] | NA [NA to NA] — Result is positive but not quantifiable | 160 [80 to 1280]

11. Secondary Outcome: Summary of Serum Concentrations (ug/mL) of MEDI6570
Description: MEDI6570 concentrations as measured in serum during the intervention and follow-up periods
Time Frame: From baseline to Day 325/Day 405
Population: All subjects who received ≥ 1 dose of MEDI6570 and have ≥ 1 one post dose evaluable MEDI6570 serum concentration will be included in the PK population. Subjects will be analysed according to the actual treatment they received. The pk data was analysed only for 50 mg, 150mg and 400mg groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg
Number analyzed (Participants) | 38 | 129 | 117
ug/mL
  Baseline | NA (NA) — All subjects had values below limit of quantification (LLOQ) | NA (NA) — All subjects had values below limit of quantification (LLOQ) | NA (NA) — All subjects had values below limit of quantification (LLOQ)
  Day 10: number analyzed (Participants) | 37 | 123 | 111
  Day 10 | 2.3126 (101.5) | 7.0296 (125.9) | 20.4472 (37.2)
  Day 29: number analyzed (Participants) | 37 | 122 | 113
  Day 29 | 0.6154 (170.7) | 3.4641 (103.2) | 9.5328 (115.4)
  Day 57: number analyzed (Participants) | 34 | 124 | 107
  Day 57 | 0.7622 (235.5) | 4.3897 (145.9) | 15.0108 (50.3)
  Day 85: number analyzed (Participants) | 22 | 33 | 85
  Day 85 | 1.1353 (217.3) | 6.4317 (62.0) | 10.8714 (608.2)
  Day 113: number analyzed (Participants) | 34 | 117 | 101
  Day 113 | 1.0084 (176.7) | 5.4403 (120.1) | 15.5611 (77.1)
  Day 122: number analyzed (Participants) | 15 | 18 | 14
  Day 122 | 4.6703 (37.0) | 8.1229 (792.0) | 28.1805 (168.8)
  Day 141: number analyzed (Participants) | 19 | 24 | 11
  Day 141 | 1.4191 (129.5) | 8.0736 (47.2) | 10.4080 (647.5)
  Day 169: number analyzed (Participants) | 17 | 101 | 97
  Day 169 | 0.8016 (171.6) | 5.2865 (163.4) | 15.9449 (145.9)
  Day 197: number analyzed (Participants) | 0 | 0 | 1
  Day 197 |  |  | NA (NA) — Not calculable. only 1 patient attend on Day 197 in this group
  Day 225: number analyzed (Participants) | 6 | 8 | 0
  Day 225 | 2.2469 (86.3) | 3.6384 (633.4) |
  Day 253: number analyzed (Participants) | 32 | 121 | 108
  Day 253 | 0.7253 (288.4) | 5.6832 (136.0) | 14.9944 (173.4)
  Day 325/Day 405: number analyzed (Participants) | 27 | 108 | 97
  Day 325/Day 405 | NA (NA) — All subjects had values below limit of quantification (LLOQ) | NA (NA) — All subjects had values below limit of quantification (LLOQ) | 0.5955 (720.6)

12. Secondary Outcome: Number of Participants With Adverse Events in Any Category
Description: To assess the safety and tolerability of MEDI6570 compared with placebo
Time Frame: During study follow-up (from day 1 to day 325)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- MEDI6570 Total: Participants received MEDI6570 50 mg or 150 mg or 400 mg every 4 weeks for 32 weeks
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | MEDI6570 Total | Placebo
Number analyzed (Participants) | 39 | 129 | 126 | 294 | 126
Participants
  Any AEs | 26 | 87 | 79 | 192 | 65
  Any AEs with outcome of death | 0 | 1 | 1 | 2 | 0
  Any SAE (including events with outcome of death) | 4 | 17 | 10 | 31 | 13
  Any AE leading to treatment discontinuation | 1 | 0 | 2 | 3 | 3
  Any AE leading to withdrawal from study | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Most Common Adverse Events (Frequency > 5%)
Description: To assess the safety and tolerability of MEDI6570 compared with placebo
Time Frame: During study follow-up (from day 1 to day 325)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | MEDI6570 Total | Placebo
Number analyzed (Participants) | 39 | 129 | 126 | 294 | 126
Participants
  Participants with any AE | 16 | 35 | 38 | 89 | 26
  COVID-19 | 3 | 8 | 17 | 28 | 6
  Hypertension | 2 | 4 | 9 | 15 | 9
  Non-cardiac chest pain | 3 | 5 | 6 | 14 | 4
  Dyspnoea | 2 | 3 | 4 | 9 | 3
  Hypotension | 2 | 1 | 4 | 7 | 1
  Angina pectoris | 2 | 10 | 3 | 15 | 6
  Pyrexia | 2 | 1 | 3 | 6 | 1
  Diarrhoea | 2 | 5 | 2 | 9 | 4
  Epistaxis | 2 | 1 | 2 | 5 | 1
  Influenza | 2 | 4 | 2 | 8 | 1
  Nausea | 2 | 1 | 1 | 4 | 1
  Pain in extremity | 2 | 1 | 1 | 4 | 1

14. Secondary Outcome: Vital Signs (Change in Systolic and Diastolic Blood Pressure From Baseline) Over Time
Description: To assess the safety and tolerability of MEDI6570 compared with placebo
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | Placebo
Number analyzed (Participants) | 39 | 129 | 126 | 126
mmHg
  Systolic blood pressure Day 10: number analyzed (Participants) | 37 | 125 | 120 | 121
  Systolic blood pressure Day 10 | 0.3 (9.9) | 0.9 (12.7) | -1.4 (13.0) | 0.4 (12.8)
  Systolic blood pressure Day 29: number analyzed (Participants) | 38 | 124 | 122 | 122
  Systolic blood pressure Day 29 | -0.7 (10.8) | -1.1 (14.6) | -1.5 (11.9) | -1.3 (12.6)
  Systolic blood pressure Day 57: number analyzed (Participants) | 34 | 126 | 116 | 119
  Systolic blood pressure Day 57 | 1.4 (11.6) | 0.7 (14.1) | -1.6 (12.3) | -0.1 (12.8)
  Systolic blood pressure Day 85: number analyzed (Participants) | 32 | 123 | 119 | 116
  Systolic blood pressure Day 85 | 0.7 (10.2) | 1.5 (13.8) | -1.2 (12.7) | -0.5 (14.9)
  Systolic blood pressure Day 113: number analyzed (Participants) | 34 | 119 | 113 | 114
  Systolic blood pressure Day 113 | -0.6 (10.6) | 1.3 (15.2) | 0.2 (13.7) | 0.6 (13.1)
  Systolic blood pressure Day 122: number analyzed (Participants) | 15 | 22 | 22 | 16
  Systolic blood pressure Day 122 | 1.6 (16.4) | -4.0 (15.5) | -2.0 (13.8) | 7.8 (17.1)
  Systolic blood pressure Day 141: number analyzed (Participants) | 35 | 119 | 117 | 112
  Systolic blood pressure Day 141 | 0.7 (15.0) | -0.2 (14.1) | -0.2 (14.1) | 0.8 (13.3)
  Systolic blood pressure Day 169: number analyzed (Participants) | 30 | 121 | 115 | 110
  Systolic blood pressure Day 169 | 1.2 (13.4) | 1.5 (12.5) | -0.3 (14.9) | 0.5 (14.5)
  Systolic blood pressure Day 197: number analyzed (Participants) | 33 | 118 | 116 | 109
  Systolic blood pressure Day 197 | 0.7 (15.8) | 0.6 (14.0) | -3.6 (13.5) | -0.4 (13.6)
  Systolic blood pressure Day 225: number analyzed (Participants) | 35 | 115 | 112 | 110
  Systolic blood pressure Day 225 | 2.8 (14.3) | 1.7 (14.8) | -0.6 (15.1) | -0.3 (14.7)
  Systolic blood pressure Day 253: number analyzed (Participants) | 36 | 123 | 116 | 114
  Systolic blood pressure Day 253 | -1.8 (15.5) | 0.7 (14.4) | -0.9 (15.6) | 0.2 (14.5)
  Systolic blood pressure Day 325/405: number analyzed (Participants) | 29 | 112 | 104 | 99
  Systolic blood pressure Day 325/405 | -1.8 (12.8) | 0.7 (14.1) | -2.5 (14.7) | 0.1 (16.0)
  Diastolic blood pressure Day 10: number analyzed (Participants) | 37 | 125 | 120 | 121
  Diastolic blood pressure Day 10 | -0.2 (6.0) | 0.6 (8.5) | -0.3 (8.4) | -0.4 (8.7)
  Diastolic blood pressure Day 29: number analyzed (Participants) | 38 | 124 | 122 | 122
  Diastolic blood pressure Day 29 | 0.3 (8.5) | -1.3 (8.7) | -1.1 (9.7) | -1.3 (9.1)
  Diastolic blood pressure Day 57: number analyzed (Participants) | 34 | 126 | 116 | 119
  Diastolic blood pressure Day 57 | -1.1 (8.5) | -0.5 (8.4) | -0.9 (8.9) | -0.4 (8.5)
  Diastolic blood pressure Day 85: number analyzed (Participants) | 32 | 123 | 119 | 116
  Diastolic blood pressure Day 85 | -0.1 (9.0) | -0.5 (10.5) | -0.9 (8.9) | -0.6 (9.2)
  Diastolic blood pressure Day 113: number analyzed (Participants) | 34 | 119 | 113 | 114
  Diastolic blood pressure Day 113 | -0.3 (8.5) | 0.1 (9.4) | -0.5 (8.9) | 1.0 (9.1)
  Diastolic blood pressure Day 122: number analyzed (Participants) | 15 | 22 | 22 | 16
  Diastolic blood pressure Day 122 | -3.7 (10.4) | -3.9 (8.0) | -2.0 (7.5) | 4.1 (12.3)
  Diastolic blood pressure Day 141: number analyzed (Participants) | 35 | 119 | 117 | 112
  Diastolic blood pressure Day 141 | -1.5 (8.4) | -1.1 (9.6) | -0.3 (8.5) | 0.2 (7.9)
  Diastolic blood pressure Day 169: number analyzed (Participants) | 30 | 121 | 115 | 110
  Diastolic blood pressure Day 169 | -0.4 (9.5) | -0.3 (9.2) | -0.8 (9.0) | -0.4 (9.2)
  Diastolic blood pressure Day 197: number analyzed (Participants) | 33 | 118 | 116 | 109
  Diastolic blood pressure Day 197 | -1.6 (7.7) | 0.0 (9.5) | -2.0 (9.8) | -0.3 (9.0)
  Diastolic blood pressure Day 225: number analyzed (Participants) | 35 | 115 | 112 | 110
  Diastolic blood pressure Day 225 | 0.4 (9.5) | -1.6 (9.8) | -0.9 (8.8) | -0.8 (8.4)
  Diastolic blood pressure Day 253: number analyzed (Participants) | 36 | 123 | 116 | 114
  Diastolic blood pressure Day 253 | -3.7 (7.9) | -0.1 (10.7) | -1.0 (9.9) | -0.4 (9.3)
  Diastolic blood pressure Day 325/405: number analyzed (Participants) | 29 | 112 | 104 | 99
  Diastolic blood pressure Day 325/405 | -1.8 (8.5) | -0.5 (9.1) | -1.5 (10.3) | -0.7 (9.8)

15. Secondary Outcome: Vital Signs (Change in Heart Rate From Baseline) Variables Over Time
Description: To assess the safety and tolerability of MEDI6570 compared with placebo
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | Placebo
Number analyzed (Participants) | 39 | 129 | 126 | 126
beats/min
  Heart rate Day 10: number analyzed (Participants) | 37 | 125 | 120 | 121
  Heart rate Day 10 | 0.4 (9.4) | 0.6 (8.0) | 0.4 (6.9) | -0.6 (8.6)
  Heart rate Day 29: number analyzed (Participants) | 38 | 124 | 122 | 122
  Heart rate Day 29 | -0.5 (11.4) | 0.7 (8.3) | 1.3 (8.2) | -1.1 (8.5)
  Heart rate Day 57: number analyzed (Participants) | 34 | 126 | 116 | 119
  Heart rate Day 57 | -2.1 (11.0) | 0.9 (8.9) | 2.5 (9.7) | 1.1 (11.1)
  Heart rate Day 85: number analyzed (Participants) | 32 | 123 | 119 | 116
  Heart rate Day 85 | -3.3 (9.4) | 1.0 (9.2) | 2.3 (8.3) | 1.3 (10.4)
  Heart rate Day 113: number analyzed (Participants) | 34 | 119 | 113 | 114
  Heart rate Day 113 | -1.8 (9.8) | 0.5 (10.1) | 0.2 (8.7) | 0.2 (10.7)
  Heart rate Day 122: number analyzed (Participants) | 15 | 22 | 22 | 16
  Heart rate Day 122 | -3.3 (10.8) | -1.2 (13.4) | -1.3 (7.6) | 0.7 (16.0)
  Heart rate Day 141: number analyzed (Participants) | 35 | 119 | 117 | 112
  Heart rate Day 141 | -1.3 (10.4) | 0.8 (9.2) | 2.0 (9.4) | 2.2 (10.4)
  Heart rate Day 169: number analyzed (Participants) | 30 | 121 | 115 | 110
  Heart rate Day 169 | 0.7 (10.1) | 0.5 (11.0) | 3.0 (8.8) | 1.5 (9.7)
  Heart rate Day 197: number analyzed (Participants) | 33 | 118 | 116 | 109
  Heart rate Day 197 | 2.1 (12.5) | 2.3 (9.8) | 1.7 (9.5) | 1.8 (10.4)
  Heart rate Day 225: number analyzed (Participants) | 35 | 115 | 112 | 110
  Heart rate Day 225 | 0.9 (10.0) | 1.2 (11.0) | 2.5 (10.1) | 1.8 (10.4)
  Heart rate Day 253: number analyzed (Participants) | 36 | 122 | 116 | 114
  Heart rate Day 253 | -0.8 (12.2) | 0.2 (11.0) | 2.1 (10.0) | 0.4 (9.4)
  Heart rate Day 325/405: number analyzed (Participants) | 29 | 112 | 104 | 99
  Heart rate Day 325/405 | 0.5 (10.4) | 1.3 (9.8) | 1.9 (9.4) | 0.7 (9.9)

16. Secondary Outcome: Vital Signs (Change of Weight From Baseline to Day 325/405 )
Description: To assess the safety and tolerability of MEDI6570 compared with placebo
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | Placebo
Number analyzed (Participants) | 39 | 129 | 126 | 126
kg | 0.316 (4.550) | 1.445 (4.863) | 1.078 (4.714) | 0.786 (5.348)

ADVERSE EVENTS:
Time Frame: During study follow-up (from day 1 to day 325/405). Day 325/405: for participants who completed the study under CSP Amendment 1 & 2, the end of study visits were Day 405 and Day 325, respectively.
Description: Subjects initially randomized to the 250 mg group switched dose to 400 mg following CSP amendment 1 and were analysed according to the 400 mg group.
Arm/Group | MEDI6570 50 mg | MEDI6570 150 mg | MEDI6570 400 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 1/129 | 1/126 | 0/126
Serious Adverse Events (participants affected / at risk) | 4/39 | 17/129 | 10/126 | 13/126
Other Adverse Events (participants affected / at risk) | 15/39 | 33/129 | 37/126 | 23/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI6570 50 mg (N=39) | MEDI6570 150 mg (N=129) | MEDI6570 400 mg (N=126) | Placebo (N=126)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Omental necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — 8 Subjects initially randomized to the 250 mg group switched dose to 400 mg following CSP amendment 1 and were analysed according to the 400 mg group.
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stag horn calculus (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — 8 Subjects initially randomized to the 250 mg group switched dose to 400 mg following CSP amendment 1 and were analysed according to the 400 mg group.
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI6570 50 mg (N=39) | MEDI6570 150 mg (N=129) | MEDI6570 400 mg (N=126) | Placebo (N=126)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (5) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 5 (5) | 6 (8) | 4 (4)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 3 (4) | 1 (1)
Covid-19 (Infections and infestations) | 2 (2) | 8 (8) | 16 (17) | 6 (6) — 8 Subjects initially randomized to the 250 mg group switched dose to 400 mg following CSP amendment 1 and were analysed according to the 400 mg group.
Angina pectoris (Cardiac disorders) | 1 (1) | 7 (7) | 3 (4) | 4 (4)
Influenza (Infections and infestations) | 2 (2) | 4 (4) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 4 (5) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (4) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 4 (5) | 9 (9) | 9 (9)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 4 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the sponsor for review before submission.

DOCUMENTS (2):
  • Study Protocol (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT04610892/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT04610892/SAP_001.pdf